CLINICAL TRIAL: NCT05619354
Title: Validity and Reliability of the Dutch Version of the Headache Disability Inventory (HDI) Questionnaire
Brief Title: Validity and Reliability of the Dutch HDI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2022-0312
Record Dates: First submitted 2022-11-07; First posted 2022-11-16 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Headache; Headache Disorders; Neck Pain; Cervical Pain
MeSH Terms: conditions — Headache; Headache Disorders; Neck Pain | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with headache: Individuals with primary or secondary headache forms.
  The Headache Disability Index will be applied:
  In the translation phase:
  1. Complete and assess the Dutch translation of the HDI questionnaire. The questionnaire and its evaluation can be completed online. If desired, the questionnaire can also be completed on paper, whereby the questions can be asked orally by a researcher.
     OR
     In the validation phase:
  2. To complete the Dutch questionnaire, in combination with other questionnaires (RAND-36 questionnaire and HIT-6 questionnaire).The questionnaires can be completed online. If desired, the questionnaires can also be completed on paper. Afterwards participants will be asked to complete the HDI questionnaire again after 1 month.
  Interventions: Other: Survey study

INTERVENTIONS:
Other: Survey study — Participants will be asked to complete and evaluate the Dutch version of the Headache Disability Index. Validity (face validity, content validity, convergent validity with the RAND-36 and HIT-6) will be determined. Second, internal consistency and test-retest reliability will be evaluated.

SUMMARY:
The aim of our study is to investigate the validity and reliability of Dutch version of the Henry Ford Hospital Headache Disability Questionnaire (HDI).

DETAILED DESCRIPTION:
There is only a limited number of questionnaires that map headache-related disability.

To gain a better understanding of the emotional and functional effects of headaches on the patient's well-being, an English questionnaire already exists: the Henry Ford Headache Disability Index (HDI). The purpose of the HDI is to map headache related disabiltiy. This 25-item questionnaire focusses on two categories; there are 13 questions in the field of emotional effects and 12 questions on functional effects of headache complaints.

Advantage: This questionnaire can be used for all headache patients, in contrast to many questionnaires that can only be used for migraine patients. (eg MIDAS, Migraine ACT, ID Migraine...) The questionnaire contains more items than the Headache Impact Test (HIT-6), consisting of 6 items. The questions are very specifically aimed at headaches and can also be used to further inquire about the anamnesis after completing the questionnaire.

Problem statement: There is no validated Dutch version yet.

Objective: to translate and validate a Dutch version of the HDI. About 250 patients with chronic headache will be recruited to determine the validity (face validity, content validity, convergent validity with the RAND-36 and HIT-6). In addition, internal consistency and short- and long-term test and retest reliability will be evaluated using the intraclass correlation coefficient (ICC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary or secondary headache, diagnosed by a neurologist according to the ICHD-3 classification.
* At least 1 day of headache in the previous month.
* Native Dutch speaking participants

Exclusion Criteria:

* All other headache types not classified by the ICHD-3 as primary or secondary headache.
* Secondary headache in combination with underlying pathological situations (infection, trauma, tumors, brain haemorrhages) or severe psychotic or mental dysfunctions or substance use/withdrawal symptoms.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of particants with primary and secondary headaches.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Headache Disability Index | 15 minutes
  Headache Disability Index evaluates the effects of headache on quality of life and disability

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Cagnie, Prof. Dr., Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - University Hospital Ghent, Ghent, Oost-Vlaanderen
  - Universiteit Gent, Ghent

IPD SHARING:
Plan to Share IPD: No